CLINICAL TRIAL: NCT00355524
Title: A Phase II, Open-label Trial, to Investigate Pharmacokinetics, Safety, Tolerability and Antiviral Activity of TMC114/Rtv b.i.d in Treatment-Experienced HIV-1 Infected Children and Adolescents
Brief Title: A Phase 2 Study to Evaluate Pharmacokinetics, Safety and Efficacy of TMC114/Ritonavir (Rtv) in Human Immunodeficiency Virus (HIV)-1 Infected Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002797; TMC114-C212
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: HIV-1; HIV Infections
Keywords: HIV-1; Darunavir; Ritonavir; TMC114
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group A with >= 20 kg to < 30 kg body weight (Experimental): 300 milligram (mg) of TMC114 tablet with 50 mg (which is equivalent to 0.625 milliliter [mL]) of ritonavir liquid (80 milligram/milliliter [mg/ml]) will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir
- Group A with >= 30 kg to < 40 kg body weight (Experimental): 300 mg of TMC114 tablet with 50 mg (which is equivalent to 0.625 milliliter [mL]) of ritonavir liquid (80 milligram/milliliter [mg/ml]) will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir
- Group A with >= 40 kg to < 50 kg body weight (Experimental): 450 mg of TMC114 tablet with 100 mg of ritonavir capsule will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir
- Group B with >= 20 kg to < 30 kg body weight (Experimental): 375 mg of TMC114 tablet with 50 mg (which is equivalent to 0.625 mL) of ritonavir liquid (80 mg/mL) will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir
- Group B with >= 30 kg to < 40 kg body weight (Experimental): 450 mg of TMC114 tablet with 60 mg (which is equivalent to 0.75 mL) of ritonavir liquid (80 mg/mL) will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir
- Group B with >= 40 kg to < 50 kg body weight (Experimental): 600 mg of TMC114 tablet with 100 mg of ritonavir capsule will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir
- Participants with >= 50 kg body weight (Experimental): 600 mg of TMC114 tablet with 100 mg of ritonavir capsule will be administered orally twice daily.
  Interventions: Drug: TMC114; Drug: Ritonavir

INTERVENTIONS:
Drug: TMC114 — TMC114 will be administered as oral tablets (75 milligram [mg] or 300 mg) twice daily at a dose ranging from 300-600 mg up to 48 weeks.
  Other Names: Darunavir
Drug: Ritonavir — Ritonavir will be administered as oral capsules (100 mg) or liquid (80 mg/mL) twice daily at a dose ranging from 50 mg (0.625 mL)-100 mg up to 48 weeks.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time), safety, tolerability and antiviral activity to support dose recommendations of TMC114 with ritonavir and other antiretroviral agents in treatment-experienced, human immunodeficiency virus (HIV)-1 infected children and adolescents.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) and randomized (study drug assigned by chance) study to evaluate pharmacokinetics, safety, tolerability, efficacy, antiviral activity, immunology and resistance characteristics of TMC114 with ritonavir in treatment-experienced, HIV-1 infected children and adolescent participants. The study consists of 3 periods: Screening period (maximum 4 weeks); Treatment period (maximum 48 weeks); and Follow-up period (4 weeks). The Treatment period consists of two parts: Part-1 for pediatric dose selection and Part-2 for the recommendation of pediatric or adult dose. Part-1 was further divided into two groups: Group A with adult equivalent dose of TMC114 with ritonavir twice daily and Group B with 20-33 percent higher dose of TMC114 with ritonavir twice daily. The recommended dose will be selected based on short-term safety, tolerability, antiviral activity and pharmacokinetics at Week 2. Once selected, all Part-1 participants who will not be on the selected dose will be switched to the selected dose at their next visit and will continue the study up to 48 weeks in Part-2. Participants with less than or equal to 18 years at Week 48 visit, and continued to benefit from treatment with TMC114 and will be living in a country where TMC114 pediatric use is not yet part of the label, will have the opportunity to roll-over to the extension phase where they will continue to receive TMC114/ritonavir until the participant became 18 years and TMC114 will be available through the local Health Care Systems or until TMC114 is indicated for use in pediatrics. Efficacy will primarily be evaluated by virologic response. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented human immunodeficiency virus (HIV)-1 infection failing their current antiretroviral therapy
* Body weight for Part 1: greater than or equal to 20 Kilogram (kg) but less than 50 kg and body weight for Part 2: greater than or equal to 50 kg and from greater than or equal to 20 but less than 50 kg after pediatric dose selection
* Able to swallow the TMC114 tablet formulations, the ritonavir capsule formulation, and to tolerate the ritonavir liquid formulation
* Stable cluster of differentiation 4 (CD4+) percentage; that is no more than 5 percent decrease in CD4+ percentage between the Screening visit and the last available CD4+ measurement
* Female participants who are sexually active and able to become pregnant must use a safe and effective birth control method

Exclusion Criteria:

* For Part 1: Use of the non-nucleoside analogue reverse transcriptase inhibitor (NNRTI) efavirenz as part of the current regimen was not allowed and for Part 2: Use of efavirenz as part of the current regimen was allowed and use of any antiretroviral and non-antiretroviral investigational agents within 30 days prior to screening
* Presence of any currently active acquired immune deficiency syndrome (AIDS) defining illness (Category C conditions according to the Centers for Disease Control [CDC] Classification System for HIV Infection 1993 or according to the 1994 revised CDC Classification System for HIV infection in children less than 13 years of age)
* Pregnant or breastfeeding female participants
* Previous allergy or hypersensitivity to any excipients of the investigational medication (TMC114) or ritonavir
* Any Grade 3 or 4 toxicity as defined by the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading scale

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time of Administration to 12 hours After Dosing (AUC 0-12h) - Part 1 | Week 2
  The Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Predose Plasma Concentration (C0) - Part 1 | Week 2
  The C0 is the predose plasma concentration.
Maximum Observed Plasma Concentration (Cmax) - Part 1 | Week 2
  The Cmax is the maximum observed plasma concentration.
Recommended Dose of TMC114 per Body Weight | Week 2
  The recommended dose of TMC114 will be determined in participants with a body weight: greater than and equal to 20 Kilogram (kg) to less than 30 kg; greater than and equal to 30 kg to less than 40 kg; and greater than 40 kg.
Change From Baseline in Plasma Viral Load at Week 2 - Part 1 | Baseline and Week 2
  Plasma viral load levels will be determined using Roche amplicor human immunodeficiency virus (HIV)-1 monitor test (Version 1.5).
Change From Baseline in Plasma Viral Load at Week 24- Part 2 | Baseline and Week 24
  Plasma viral load levels will be determined using Roche amplicor HIV-1 monitor test (Version 1.5).
Number of Participants With Adverse Events | Week 2
  Adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product and which does not necessarily have a causal relationship with the treatment.
Number of Participants With Adverse Events | Week 24
  Adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product and which does not necessarily have a causal relationship with the treatment.

SECONDARY OUTCOMES:
Change From Baseline in Plasma Viral Load at Week 48 - Part 2 | Baseline and Week 48
  Plasma viral load levels will be determined using Roche amplicor HIV-1 monitor test (Version 1.5).
Change from Baseline in Cluster of Differentiation 4 (CD4+) cell count - Part 2 | Baseline and Week 48
  The immunologic change will be determined by changes in CD4+ cell count.
Number of Participants With Resistance - Part 2 | Week 48
  Resistance will be determined by viral phenotype and genotype determinations, which will be performed by Virco BVBA, by means of the antivirogram and Virco type HIV-1 respectively. Resistance determinations will only be generated if the viral load is greater than 1000 HIV-1 RNA copies/milliliter.
Area Under the Plasma Concentration-Time Curve From Time of Administration to 12 hours After Dosing (AUC 0-12h) - Part 2 | Week 48
  The Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Predose Plasma Concentration (C0) - Part 2 | Week 48
  The C0 is the predose plasma concentration.
Oral Clearance (CL/F) - Part 2 | Week 48
  The CL/F is the oral clearance; that is clearance based on oral bioavailability.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (22):
- United States (7):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
- Buenos Aires, Argentina
- Brazil (4):
  - Belo Horizonte
  - Nova Iguaçu
  - Ribeirão Preto
  - Rio de Janeiro
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Paris, France
- Romania (2):
  - Bucharest
  - Constanța
- South Africa (3):
  - Cape Town Cape
  - Durban
  - Johannesburg Gauteng
- Spain (2):
  - Esplugues de Llobregat
  - Madrid

REFERENCES:
- [Result] Blanche S, Bologna R, Cahn P, Rugina S, Flynn P, Fortuny C, Vis P, Sekar V, van Baelen B, Dierynck I, Spinosa-Guzman S. Pharmacokinetics, safety and efficacy of darunavir/ritonavir in treatment-experienced children and adolescents. AIDS. 2009 Sep 24;23(15):2005-13. doi: 10.1097/QAD.0b013e328330abaa. PMID 19724191
- See also: A Phase II, Open-label Trial, to Investigate Pharmacokinetics, Safety, Tolerability and Antiviral Activity of TMC114/rtv b.i.d in Treatment-Experienced HIV-1 Infected Children and Adolescents — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=987&filename=CR002797_CSR.pdf